CLINICAL TRIAL: NCT06714981
Title: A Comparison of Opioid-Free Anesthesia (OFA) and Standard Fentanyl-based General Anesthesia in Patients with Morbid Obesity Undergoing Laparoscopic Bariatric Surgery
Brief Title: Hemodynamics Stability During Opioid Free Anesthesia for Patients with Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Lodz (Other)
Responsible Party: Principal Investigator, Tomasz Gaszynski, professor of anesthesia, Medical University of Lodz
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RNN/60/16/KE
Record Dates: First submitted 2024-11-25; First posted 2024-12-04 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-11

CONDITIONS: Obesity; General Anesthesia; Opioid Free Anaesthesia
Keywords: general anesthesia; Opioid-Free Anesthesia; obesity; fentanyl; hemodynamics
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- opioid free anesthesia (Experimental): patients received opioid free anesthesia
  Interventions: Drug: Opioid Free Anaesthesia
- opioid based anesthesia (Active Comparator): patients received opioid based anesthesia
  Interventions: Drug: Opioid based Anesthesia

INTERVENTIONS:
Drug: Opioid Free Anaesthesia — patients received opioid free anesthesia
  Arms: opioid free anesthesia
Drug: Opioid based Anesthesia — patients received opioid based anesthesia
  Arms: opioid based anesthesia

SUMMARY:
The study evaluated the impact of Opioid-Free Anesthesia (OFA) and Fentanyl Anesthesia (FNT) on the hemodynamics of the circulatory system (HR, esCCO, esCCI, esSVI, BP: SYS, DIA, MEAN) in obese patients with a BMI > 40 undregoing laparoscopic bariatric surgery. Patients in the OFA group were anesthetized as follows: before induction: ketamine 0.15 mg/kg (corrected body weight), lidocaine 1-1.5 mg/kg (corrected body weight) slow infusion, magnesium sulfate 30-50 mg/kg (corrected body weight), dexamethasone 8 mg, paracetamol 2.0g. Maintenance: continuous infusion of ketamine 0.125-0.25 mg/kg/h (corrected body weight), lidocaine 1.5-3 mg/kg/h (corrected body weight), magnesium sulfate 10 mg/kg/min (corrected body weight), and rocuronium bromide 1.25 µg/kg/min (corrected body weight) were used. Patients in the FNT group were anesthetized as follows: before induction: fentanyl 1.5-3 µg/kg (corrected body weight) iv, preoxygenation with 100% oxygen for 3 minutes, propofol 2.5 mg/kg (actual body weight) and following confirmation of mask ventilation, rocuronium bromide 0.6 mg/kg (actual body weight) bolus. After achieving full neuromuscular blockade, the patient was intubated and connected to the anesthesia machine and ventilated with 1-1.5 MAC desflurane.

DETAILED DESCRIPTION:
Adult patients (over 18 years old) with a BMI ≥ 40, ASA ≤ II, qualified for elective bariatric surgery under general anesthesia with endotracheal intubation, who provided informed, voluntary consent to participate in the study, were included. Patients with BMI < 40, ASA III and above, heart failure, arrhythmias (especially bradyarrhythmia), hypovolemia, shock, unstable coronary artery disease, autonomic neuropathy with orthostatic hypotension, with a history of allergic reactions, pregnancy, indications for urgent surgical intervention, or those who did not consent to participate in the study, were excluded. Patients' weight, height, and BMI were measured. All obtained data were anonymized.

After transporting the patient to the operating room, the envelope was opened, and the patient was assigned to either the OFA or FNT anesthesia group.

Patients in the OFA group were anesthetized as follows: before induction: ketamine 0.15 mg/kg (corrected body weight), lidocaine 1-1.5 mg/kg (corrected body weight) slow infusion, magnesium sulfate 30-50 mg/kg (corrected body weight), dexamethasone 8 mg, paracetamol 2.0g. Induction: after three minutes of preoxygenation with 100% oxygen, propofol 2.5 mg/kg (actual body weight) was administered. Following confirmation of mask ventilation, rocuronium bromide 0.6 mg/kg (actual body weight) was given. Bag-mask ventilation with 100% oxygen continued for 3 minutes. After achieving full neuromuscular blockade, confirmed by the loss of all four responses using a peripheral nerve stimulator, the patient was intubated and connected to the anesthesia machine and ventilated with 1-1.5 MAC sevoflurane. Maintenance: ketamine 0.125-0.25 mg/kg/h (corrected body weight), lidocaine 1.5-3 mg/kg/h (corrected body weight), magnesium sulfate 10 mg/kg/min (corrected body weight), and rocuronium bromide 1.25 µg/kg/min (corrected body weight) were used. After surgery, neuromuscular blockade was reversed with sugammadex at 2-4 mg/kg (corrected body weight). The patients were also administered ephedrine in case of hypotension, atropine for bradycardia, and beta-blockers for tachycardia and hypertension.

Patients in the FNT group were anesthetized as follows: before induction: fentanyl 1.5-3 µg/kg (corrected body weight) iv, preoxygenation with 100% oxygen for 3 minutes, propofol 2.5 mg/kg (actual body weight) and following confirmation of mask ventilation, rocuronium bromide 0.6 mg/kg (actual body weight) bolus. Bag-mask ventilation with 100% oxygen and 2% inhaled sevoflurane continued for 3 minutes. After achieving full neuromuscular blockade, the patient was intubated and connected to the anesthesia machine and ventilated with 1-1.5 MAC desflurane. Maintenance dose for fentanyl was 0.003-0.006 µg/kg/min (corrected body weight) and rocuronium bromide 1.25 µg/kg/min (corrected body weight) were used. After surgery, neuromuscular blockade was reversed with sugammadex at 2-4 mg/kg (corrected body weight).

During induction, patients were positioned supine with the head and torso elevated at a 25-degree angle on a positioning pad. Anesthetic monitoring included HR, NIPC-SYS, NIPC-MEAN, NIPC-DIA, SpO2, esCCO, esCCI, and esSVI using the Vismo monitor and EtCO2.

Hemodynamic parameters (esCCO, esCCI, esSVI, NIPC-SYS, NIPC-MEAN, NIPC-DIA, HR) were measured before induction (T0) and then at 10-minute intervals after intubation and connection to the anesthesia machine (from T1 to T10).

The objective of the study is to compare the impact of OFA on hemodynamic parameters measured by non-invasive technique: esCCO, esCCI, esSVI, NIPC-SYS, NIPC-MEAN, NIPC-DIA, HR, in obese patients with BMI > 40, with those obtained during the commonly used FNT anesthesia.

ELIGIBILITY:
Inclusion Criteria:

- obese patients with a BMI > 40 kg/m2 undergoing elective laparoscopic bariatric surgery

Exclusion Criteria:

* lack of consent
* emergency operation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-01-02 (Actual); Primary Completion 2023-01-02 (Actual); Study Completion 2023-06-02 (Actual)

PRIMARY OUTCOMES:
hemodynamic stability, cardiac output | before induction (T0) and then at 10-minute intervals after intubation and connection to the anesthesia machine (from T1 to T10)
  Hemodynamic parameters (esCCO - cardiac output l/min) were measured using Visimo monitor.
hemodynamic stability esCCI - cardiac index | before induction (T0) and then at 10-minute intervals after intubation and connection to the anesthesia machine (from T1 to T10)
  Cardiac index esCCI - l/m2 was measured using Visimo monitor.
hemodynamic stability esSVI | before induction (T0) and then at 10-minute intervals after intubation and connection to the anesthesia machine (from T1 to T10)
  Stroke voulme esSVI - l were measured using Visimo monitor.
hemodynamic stability: arterial pressure NIPC-SYS, NIPC-MEAN, NIPC-DIA | before induction (T0) and then at 10-minute intervals after intubation and connection to the anesthesia machine (from T1 to T10)
  Arterial pressure NIPC-SYS, NIPC-MEAN, NIPC-DIA (mmHg) were measured using Visimo monitor.
hemodynamic stability HR - heart rate | before induction (T0) and then at 10-minute intervals after intubation and connection to the anesthesia machine (from T1 to T10)
  HR were measured using Visimo monitor.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Lodz, Lodz, Poland

IPD SHARING:
Plan to Share IPD: No